CLINICAL TRIAL: NCT06910176
Title: Confirming And Notifying Death : Blended Learning and Its Evaluation by Medical Students, an Acceptability Study"
Brief Title: Confirming And Notifying Death
Acronym: CANDELS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9304
Record Dates: First submitted 2025-03-27; First posted 2025-04-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-03

CONDITIONS: Death Records
Keywords: Notifying Death; Death Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most physicians are confronted with the death of patients during their practice, often as early as residency. It is their legal responsibility to certify a patient's death, as well as often to notify their loved ones.

Yet, these duties currently receive little or no specific training during the various cycles of medical education.

This task is not easy, however, and young professionals experience it with difficulty. Literature data show that residents are confronted with death late in their medical education and that they are insufficiently prepared when they have to perform their first death certificate. Indeed, residents report significantly correlated practical and emotional difficulties. These difficulties are notably linked to a feeling of lack of preparation through theoretical courses, a lack of familiarity with administrative procedures, and insufficient mastery of communicating with families. The highlighting of these difficulties and the desire for appropriate and respectful care for the deceased and their families, for whom the moment of announcement influences the experience of grief, call for an improvement in teaching on these topics. It is in this sense that the project was born to explore whether the creation of training, before their independent exposure to death and its announcement, i.e. at the end of the second cycle, was relevant. A prerequisite for this type of training project is indeed to question the acceptability of such an approach by students.

ELIGIBILITY:
Inclusion Criteria:

* DFASM3 student,
* At the Faculty of Medicine of Strasbourg, France, for the 2023-2024 academic year,
* Having taken the national ECOS (thus becoming an intern at the start of the following academic year in November 2024),
* Aged 18 years or older,
* Not opposed to participating in the study.
* Not having completed an internship in specialized palliative care facilities

Exclusion Criteria:

* Refused to participate in the study.
* Not having taken the national ECOS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Student having taken the national ECOS (thus becoming an intern at the start of the following academic year in November 2024),
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
To assess the acceptability of training in death certification and death notification to relatives by DFASM3 students in Strasbourg. | At 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de soins Palliatifs - CHU de Strasbourg - France, Strasbourg, France